CLINICAL TRIAL: NCT05162313
Title: Comparison Between Flow Sensor and Colourimetric Capnometer in Verifying the Correct Positioning of the Endotracheal Tube in Term and Preterm Infants
Brief Title: Flow Sensor and Colourimetric Capnometer in Verifying Tracheal Tube Positioning in Term and Preterm Infants
Acronym: FlowNET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Paolo Biban, Director, Neonatal Intensive Care Unit, Dept. Neonatal and Pediatric Critical Care, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2880CESC
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Tracheal Intubation
Keywords: tracheal intubation; tracheal tube positioning; colorimetric capnometer; flow sensor; invasive mechanical ventilation; newborn; preterm infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Simultaneous assignment, as the two methods to confirm the endotracheal tube position, namely the colorimetric capnometer and the flow sensor signal, will be evaluated simultaneously in each recruited patient.
Masking Description: Participants are newborns. The care provider will be the attending physician performing the tracheal intubation procedure as per local protocols, including the colourimetric capnometry analysis. However, he/she will remain blind and not aware of the flow sensor data until the end of the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all patients undergoing tracheal intubation procedure (Other): In current practice, the endotracheal intubation procedure includes the systematic use of the capnometer, which is immediately connected to the tube after its insertion by direct laringoscopy. Confirmation of the correct tube positioning is established by color change of the capnometer from violet to yellow. Then, the colorimetric capnometer is usually removed before connecting the endotracheal tube to the flow-sensor of the ventilator.
  For the purpose of our study, after the tube insertion the care provider will connect in line both the capnometer and the ventilator flow-sensor to the tracheal tube.
  Interventions: Device: confirmation of endotracheal tube positioning

INTERVENTIONS:
Device: confirmation of endotracheal tube positioning — After performing the tube insertion by direct laryngoscopy, videolaringoscopy or fiberoptic technique, the attending neonatologist will connect both the colorimetric capnometer and the proximal flow-sensor to the tracheal tube. If the flow sensor is not proximal but incorporated into the mechanical ventilator, the care provider will connect the capnometer only. During the procedure, the information given by the capnometer will be evaluated by the care provider performing the intubation, while the flow sensor information will be monitored only by a study investigator, who will not reveal any details to the care provider. In particular, the yellow color change by the capnometer and the presence of exhalation flow curves on the ventilator screen will be considered as confirmation of correct tracheal tube positioning, respectively.

SUMMARY:
This is a multicentre clinical trial with medical device. As currently recommended by international neonatal resuscitation guidelines, the most reliable method to verify the correct positioning of the endotracheal tube, in association with clinical signs, is the end-tidal capnometry obtained either by infrared spectroscopy or colorimetric method. The aim of the present study is to evaluate whether the flow sensor of a standard mechanical ventilator can discriminate with similar or faster times the correct positioning of the tube after a tracheal intubation attempt compared to the colorimetric capnometer, in newborns undergoing this procedure during hospitalization in the neonatal intensive care unit.

Given the importance of defining a rapid and effective method to prevent possible adverse events of incorrect endotracheal intubation, this study aims to verify whether the ventilator flow sensor can allow a reliable assessment of the correct positioning of the endotracheal tube, with timing and success rates equivalent to or better than the colorimetric capnometer.

DETAILED DESCRIPTION:
Specifically, the neonatologist performing the procedure will follow the standard procedure for tracheal intubation, which includes using a colourimetric capnometer to confirm the correct tube positioning. However, he/she will remain blind and not aware of the flow sensor signal, while a study investigator will monitor that.

The investigators will measure the percentage of responses of correct positioning of the endotracheal tube as well as the number of insufflations and the time elapsed before obtaining a signal of correct intubation by simultaneously comparing both methods and checking any differences based on the characteristics of the sample analyzed (e.g. premature infants versus term infants, elective versus emergency intubations).

ELIGIBILITY:
Inclusion Criteria:

Term and preterm infants requiring tracheal intubation within the neonatal intensive care unit, both in elective and emergency conditions.

Exclusion Criteria:

* intubation at birth
* intubation during cardiopulmonary resuscitation
* absence of informed consent by parents

Ages: 20 Minutes to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Time taken by the flow-sensor to indicate the correct or not correct positioning of the tracheal tube, compared with time taken by the colorimetric capnometer. | Immediately after the tracheal intubation attempt
  To compare the time (expressed in seconds) taken by the flow sensor and the colorimetric capnometer, respectively, to indicate the correct or not correct positioning of the tube in newborns undergoing tracheal intubation procedure during neonatal intensive care unit admission.
  The aim is to evaluate if the flow sensor of the mechanical ventilator can discriminate with similar or faster times the correct positioning of the tube during the tracheal intubation procedure compared to the colorimetric capnometer.
Number of mechanical breaths necessary to indicate the correct or not correct positioning of the tracheal tube by evaluating the flow-sensor curves and the color change of the colorimetric capnometer. | Immediately after the tracheal intubation attempt
  To compare the minimal number of mechanical breaths provided by the ventilator to indicate the correct or not correct positioning of the tube in newborns undergoing tracheal intubation procedure, either evaluating the flow-sensor curves and the color change of the colorimetric capnometer, respectively.
  The aim is to evaluate if the flow sensor of the mechanical ventilator can indicate with lower or equal number of mechanical breaths the correct positioning of the tube during tracheal intubation compared to the colorimetric capnometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy